CLINICAL TRIAL: NCT06530654
Title: Augmented Reality as a Distraction Technique in Paediatric Dental Care, Assessment of Resulting Effects on Patient Anxiety, Pain and Behaviour
Brief Title: Effect of Augmented Reality on Dental Anxiety and Pain Perception in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Istanbul Technical University (Other)
Responsible Party: Principal Investigator, Yelda Kasımoğlu, Principal investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 123S793
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Pain
Keywords: Pain Management; Anxiety; Child; Application Software Development; Augmented Reality; Human Computer Interaction
MeSH Terms: conditions — Anxiety Disorders; Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard treatment group (Active Comparator): Basic behavior orientation techniques (tell-show-do) is applied by the dentist during the treatment.
  Interventions: Behavioral: Distraction by dentist
- Cartoon movie- passive distraction group (Experimental): Children watch cartoons on a screen mounted dental unit during the treatment.
  Interventions: Behavioral: Distraction by cartoon movie
- AG-active distraction group (Experimental): A tablet will be used for AG notation. How to use AG will be shown to the pediatric patient just before the treatment. Since it is aimed to keep the verbal communication of the dentist with the child at the lowest level, a similar "tell-show-do" technique used in the control group will be digitally simulated on the AG. The instruments that the dentist will use during the procedure will be promoted on AG using animated content.
  Interventions: Behavioral: AG-active distraction group

INTERVENTIONS:
Behavioral: Distraction by dentist — Dental treatment is carried out with tell-show-do technique as a behavioural guidance technique.
  Arms: Standard treatment group
Behavioral: Distraction by cartoon movie — Dental treatment is carried out with showing cartoon movie as a passive distraction during the treatment.
  Arms: Cartoon movie- passive distraction group
Behavioral: AG-active distraction group — The active distraction group is treated and interacting with the designed application
  Arms: AG-active distraction group

SUMMARY:
The aim of this study is to reduce dental anxiety in children by using augmented reality (AG) with a special content and innovative interactive methods, to determine the level of stress experienced by patients during dental treatment and to ease the workload of dentists.

The effectiveness of augmented reality system is tested by comparing evaluation metrics of three groups of children. In the first group, the dentist carries out the treatment alone. In the second group participants watch cartoons on a screen mounted dental unit during the treatment. In the third group, dental treatment is carried out with AG. In the course of these experiments, the effects of AG on dental treatment (vital pulpotomy and dental filling) that require local anesthesia is examined in order to measure the effects of AG on the level of stress on dental treatment.

Corresponding measures are; (1) the child's anxiety; (2) the child's pain perception during local anaesthesia and treatment; (3) the child's cooperation and general behaviour. The outcomes of the child's anxiety, pain perception, cooperation and general behaviour for three groups were evaluated by statistical analysis.

DETAILED DESCRIPTION:
Dental anxiety can be seen in all age groups with frequency varying between 10-36% and can have negative impacts on patients and doctors. It may interrupt treatment or cause patients to avoid treatment altogether, potentially resulting in an increase in oral and dental health problems. Studies show it's possible to prevent dental anxiety at younger ages. Among basic behavior management techniques, dentists frequently depend on the distraction method to relieve patient anxiety. Literature suggests contemporary technological solutions are prominently used for distracting patients during or before dental procedures.

Literature shows robot-guided dental treatments can reduce anxiety. However, the high cost of robots, need for additional staff to direct the robot, and decrease in the overall interaction quality due to noise limit their use in clinical environments. Other studies suggest virtual reality (VR) for pediatric dental anxiety. Although VR has been successful in alleviating dental anxiety, a number of factors make it less preferable. Having to wear bulky glasses for interaction may cause discomfort to the patient. Physicians may find these devices impractical as their dimensions restrict the doctor's working area. Furthermore, completely isolating the patient from the clinic environment may cause additional anxiety. This study proposes an augmented reality (AR) approach to ease dental anxiety in pediatric patients. Using AR as a distraction technique, patients can still interact with virtual entities as if they're part of the real world, without having to be completely isolated from the clinical environment.

This study aims to reduce dental anxiety and pain perception in children by using an AR application both before and during treatment. Content especially prepared for dental treatment will be presented to patients using an innovative mobile AR interaction system. Patients will interact with the AR system in three stages. First, before treatment, the application will inform patients about equipment used during treatment. Patients will be able to interact with informative and entertaining virtual content superimposed on the real environment with avatars guiding them. The content and interaction are expected to relieve dental anxiety and increase the success rates in pediatric dental treatments. Second, the AR screen will act as a virtual stage mounted in a position that the patient can see comfortably during treatment. The child will be able to relate to virtual entities without being isolated from the environment, unlike in virtual reality solutions. Third, a rich and immersive interaction experience will be provided following treatment within the framework of gamification and personalization principles.

The effectiveness of the AR system will be evaluated by cross comparison with two other groups of patients. The control group will receive traditional dental treatment. The cartoon group will watch a cartoon movie during treatment. For the purposes of this study, tooth extraction and filling procedures that require local anesthesia will be applied to all three groups. Salivary cortisol, α-Amylase and Chromogranin (CHGA) levels will be compared to pulse measurements and evaluated with psychometric scales to determine the effects of AR on dental anxiety levels of pediatric patients.

It is expected that the stress and workload experienced by dentists will be reduced, and the child's dental treatment session will be made more comfortable for the dentist, patient and parent. Additionally, reduction of the need for high-cost equipment and qualified teams required within the scope of advanced behavior guidance techniques used to complete dental treatments in children whose dental anxiety and fear cannot be eliminated is one of the significant impacts of this study. This study is the first study in the world in which an AR system will be utilized in the field of dental treatment in order to reduce dental anxiety in children.

ELIGIBILITY:
Inclusion Criteria:

* Systemically and mentally healthy patients without any previous dental treatment experience,
* Children who required pulpotomy in lower primary molars under local anaesthesia.

Exclusion Criteria:

* Systemic disease,
* Mental and cognitive disorders, visual and auditory disabilities.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Child's anxiety assessment (objective) | 1 year
  In order to determine the stress levels of the children included in the study, cortisol, α-Amylase and CHGA levels in saliva will be measured

SECONDARY OUTCOMES:
Child's anxiety assessment (objective) | 1 year
  Heart rate is used to determine the anxiety levels of all treated children at certain critical moments of the treatment being. Significant differences in heart rate is compared between groups.
Child's anxiety assessment (subjective) | 1 year
  Scores on the Modified Child Dental Anxiety Scale, MCDAS(f) scale may range from 8 to 40, with scores below 19 indicating absence of state anxiety, scores higher than 19 indicating the pres- ence of state anxiety and scores higher than 31, in- dicating severe phobic disorder
Child's pain assessment (subjective) | 1 year
  The Wong-Baker Faces Pain Rating Scale is a method for someone to self-assess and effectively communicate the severity of pain they may be experiencing. The scale contains a series of six faces ranging from a happy face at 0 to indicate "no hurt" to a crying face at 10 to indicate "hurts worst.
Child's behaviour assessment (subjective) Child's pain assessment (subjective) | 1 year
  According to the The Frankl Behavior Rating Scale, the child's attitude towards treatment is divided into 4 groups and scored between 1-4 meaning: 1 point absolutely negative (child refuses treatment, strong fear and crying), 2 points negative (reluctant to accept treatment), 3 points positive (child accepts treatment, but is cowardly and timid) 4 points absolutely positive (compatible with pediatric dentist).

CONTACTS AND LOCATIONS:
Overall Officials: Elif Tuna Ince, Prof.Dr., Study Director — Department of Pedodontics, Faculty of Dentistry, Istanbul University
Locations (1):
- Istanbul University, Faculty of Dentistry, Department of Pedodontics, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No